CLINICAL TRIAL: NCT05649878
Title: Evaluation of the Bioavailability of Methylprednisolone Succinate Administered Intranasally
Brief Title: Evaluation of the Bioavailability of Methylprednisolone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edda Sciutto Conde (Other)
Responsible Party: Sponsor-Investigator, Edda Sciutto Conde, Principal Investigator, Universidad Nacional Autonoma de Mexico
Organization: Universidad Nacional Autonoma de Mexico (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE-PNO-049-F01
Record Dates: First submitted 2022-11-23; First posted 2022-12-14 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Methylprednisone Administration; Intranasal Administration; Intravenous Administration; Healthy Subjects
Keywords: methylprednisolone; intranasal; pharmacokinetics; Bioavailability

STUDY DESIGN:
Intervention Model Description: A single dose design was used, with 8 subjects under fasting conditions, two periods, two sequences, open, crossed with blocks scheme A-B and B-A, randomized, longitudinal, comparative and prospective, with a washout period of seven days between the two study sessions. The treatment groups were balanced, having an equal number of subjects who were randomly assigned to the administration sequences of the drug under study.
  MEP sodium succinate was administered intravenously (1 mL, equivalent to 62.5 mg of Methylprednisolone) or the same dose intranasally by 2 using a Mucosal Atomization Device (MAD Nasal).
  The nominal doses were similar, allowing direct pharmacokinetic comparison without dose normalization. Venous blood samples were obtained via an indwelling catheter before administration at different times. Plasma was separated and frozen at -70 °C for further analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenously MEP (Active Comparator): Single dose of MEP sodium succinate intravenously administered. MEP (equivalent to 62.5 mg of Methylprednisolone).
  Samples were obtained at 0.333, 0.50, 0.667, 0.833, 1, 1.0, 2, 3, 4, 6, 8, 10, 12 and 24 h after MEP administration.
  Interventions: Drug: Evaluation of bioavailability of methylprednisolone succinate administered intravenously
- Intranasally MEP (Active Comparator): Volunteers were randomly assigned to receive a single dose of MEP intranasally administered (equivalent to 62.5 mg of Methylprednisolone), using a Mucosal Atomization Device (MAD Nasal). Samples were obtained at 0.333, 0.50, 0.667, 0.833, 1, 1.0, 2, 3, 4, 6, 8, 10, 12 and 24 h after MEP administration.
  Interventions: Drug: Evaluation of bioavailability of methylprednisolone succinate administered intranasally

INTERVENTIONS:
Drug: Evaluation of bioavailability of methylprednisolone succinate administered intravenously — Bioavailability of methylprednisolone in healthy subjects of both genders, when administered intravenously. The nominal doses were similar, volunteers were randomly assigned to receive a single dose of MEP by IV bolus of 1.5 mL. Venous blood samples were obtained via an indwelling catheter before administration and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12 and 24 h for DXM. Plasma was separated and frozen at -70 °C for further analysis.
  Arms: Intravenously MEP
Drug: Evaluation of bioavailability of methylprednisolone succinate administered intranasally — Bioavailability of methylprednisolone in healthy subjects of both genders, when administered intranasally. Volunteers were randomly assigned to receive a single dose of MEP intranasally by using a Mucosal Atomization Device (MAD Nasal). allowing direct pharmacokinetic comparison without dose normalization. Venous blood samples were obtained via an indwelling catheter before administration and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12 and 24 h for DXM. Plasma was separated and frozen at -70 °C for further analysis.
  Arms: Intranasally MEP

SUMMARY:
This study is aimed to evaluate the bioavailability of methylprednisolone in healthy subjects of both genders, with administration intranasally versus intravenous

DETAILED DESCRIPTION:
The most important property of a drug dosage is its ability to deliver the active ingredient to the site of action in a quantity sufficient to exert the expected pharmacological effect. This ability is known as bioavailability. Methylprednisolone is a drug with wide clinical use in patients with inflammatory pathologies (infectious or non-infectious). The main routes of administration are oral and intravenous. The intranasal route could be one more effective, less invasive that would allow to obtain a faster therapeutic concentration and in greater concentration in the lungs and in the central nervous system than the intravenous route, maintaining very similar systemic concentrations to those achieved intravenously. For these reasons, it is important to know the bioavailability of methylprednisolone administered by this route in order to establish the best dosing regimen. The pilot study is of an exploratory nature (descriptive, comparative or informative), whose objective is to know the pharmacokinetic characteristics of a new route of administration of a drug in the study population to establish the pharmacokinetic parameters, and the comparison between the intranasal bioavailability against the intravenous administration by determining confidence intervals and calculating one-sided double t of Scuirmann.

Objetive: To evaluate the bioavailability of methylprednisolone in healthy subjects of both genders, with administration intranasally versus intravenous dose of 1 ml of methylprednisolone sodium succinate equivalent to 62.5 mg of methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 55 years. Clinically healthy. Body mass index between 18.0 and 27.0 Kg/m2. Negative results to detect the presence of human immunodeficiency virus [HIV], Hepatitis B [HBV], Hepatitis C [HCV) and test for detection of Syphilis (VDRL).

Subjects with negative results in tests for the detection of drugs of abuse such as: amphetamines, benzodiazepines, cocaine, methamphetamines, morphine and tetrahydro-cannabinoids.

Negative (qualitative) pregnancy test.

Exclusion Criteria:

Subjects with any condition or alteration of the nose or nasal mucosa. Subjects with a history of hypersensitivity to the study drug. Subjects with a history of cardiovascular, renal, hepatic, metabolic, gastrointestinal, neurological, endocrine, hematopoietic disorders (any type of anemia), mental illness or other organic abnormalities that could affect the pharmacokinetic study of the product under study.

Subjects who require any medication during the course of the study. Principal Investigator will not include the subject in the study. Subjects who have been hospitalized for any reason within the sixty days prior to the start of the study or who have been seriously ill within the thirty days prior to the start of the study.

Subjects who have received an investigational drug within ninety days prior to the start of the study.

Subjects who have donated or lost 450 ml or more of blood within the ninety days prior to the start of the study.

Subjects who have smoked tobacco, ingested alcohol, consumed beverages or foods containing xanthines.

Positive (qualitative) pregnancy test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability of Methylprednisolone, Intranasal Route vs. Intravenous Route | 2 weeks
  The sample size used for this exploratory study (descriptive, comparative or informative) made it possible to determine the absolute bioavailability (with informative value), for which the bioavailability was compared in the 2 types of administration: Intranasal vs. Intravenous with a sample size of 8 research subjects, even though the ANADEVA is informative, the requirements regarding type I error (alpha), type II error (beta) and a minimum difference to detect between the 2 routes of administration: intranasal vs. IV.
  The realization of the present study allowed to know the pharmacokinetic and safety parameters of the drug MEP administered by 2 different routes, as well as to determine the CVintra%

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional Autonoma de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No